CLINICAL TRIAL: NCT06144333
Title: Collection of Additional Biological Samples From Potentially COVID-19 Patients for Monitoring of Biological Parameters Carried Out as Part of the Routine
Acronym: CEB Covid-19
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CerbaXpert (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A02195-38
Record Dates: First submitted 2023-11-17; First posted 2023-11-22 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational arm (Other)
  Interventions: Diagnostic Test: RIPH2

INTERVENTIONS:
Diagnostic Test: RIPH2 — * Blood sampling by capillary
  * Swab sampling
  * Blood sampling by venous punction
  * Salivary sample, sputum, expectoration:

SUMMARY:
Patients infected with SARS-CoV-2 can present with a wide range of manifestations clinical conditions, ranging from no symptoms to serious or chronic illness. The current gold standard test for the diagnosis of COVID-19 is based on a molecular test of reverse transcription polymerase chain reaction (RT-PCR), aimed at detecting the RNA of the virus in respiratory samples such as nasopharyngeal swabs or aspirates bronchial, other methods such as antigen tests and serological detection tests IgM and IgG in response to COVID-19 viral infection, can be used for the purposes of screening in the general population.

In this context of variety of existing tests, it is important to monitor the biological parameters related to COVID-19 pathology by tracking the accuracy, specificity and sensitivity of these tests in current clinical practice.

This research is a collection of additional biological samples with minimal impact on the intake usual care of the patients concerned, for the monitoring of biological parameters carried out in routine on several reagent kits used for screening for the SARS-CoV-2 virus, in terms of sensitivity, specificity, positive and negative predictive values, for the implementation of indicators quality monitoring of these kits.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient coming for a biological analysis as part of the care for prevention, screening or monitoring of the pathogen target
* Patient able to understand the information note and give a free and informed consent, on paper or digital media
* Clinical patients:

  * Control cases (all comers or ambulatory)
  * Known positive for the pathology concerned
  * Patient hospitalized for the pathology concerned
* Pregnant or breastfeeding patient
* Dialysis patient

Exclusion Criteria:

* Patient already included in a research protocol
* Patient having received medication or treatment experimental or investigational during the last four weeks before collection
* Patient subject to a legal protection measure
* Patient affiliated with state medical aid (AME)
* Patient not affiliated to the compulsory Social Security system
* Refusal or inability to provide signed informed consent
* According to the investigator, the patient is not eligible for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7500 (Estimated)
Dates: Start 2024-12-23 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-11-23 (Estimated)

PRIMARY OUTCOMES:
Monitoring of biological parameters carried out in routine on several reagent kits used for screening for the SARS-CoV-2 virus | 24 months